CLINICAL TRIAL: NCT00597935
Title: Operations and Pelvic Muscle Training in the Management of Apical Support Loss: The OPTIMAL Trial: A Randomized Trial of Sacrospinous Ligament Fixation (SSLF) Versus Uterosacral Ligament Suspension (ULS) With and Without Perioperative Behavioral Therapy/Pelvic Muscle Training
Brief Title: Operations and Pelvic Muscle Training in the Management of Apical Support Loss: The OPTIMAL Trial
Acronym: OPTIMAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NICHD Pelvic Floor Disorders Network (Network)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 16P01; 2U01HD041249 (NIH); 2U10HD041250 (NIH); 2U10HD041261 (NIH); 2U10HD041267 (NIH); 1U10HD054136 (NIH); 1U10HD054214 (NIH); 1U10HD054215 (NIH); 1U10HD054241 (NIH)
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Pelvic Organ Prolapse (POP)
Keywords: prolapse; urinary incontinence; uterosacral vaginal vault ligament suspension; sacrospinous ligament fixation; behavioral therapy; pelvic muscle training
MeSH Terms: conditions — Pelvic Organ Prolapse; Prolapse; Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- SSLF and PMT (Experimental): Sacrospinous Ligament Fixation (SSLF) and Pelvic Muscle Training & Exercises (PMT)
  Interventions: Procedure: SSLF; Behavioral: PMT
- ULS and PMT (Experimental): Uterosacral Vaginal Vault Ligament Suspension (ULS) and Pelvic Muscle Training & Exercises (PMT)
  Interventions: Procedure: ULS; Behavioral: PMT
- SSLF without PMT (Experimental): Sacrospinous Ligament Fixation (SSLF) without Pelvic Muscle Training & Exercises (PMT)
  Interventions: Procedure: SSLF
- ULS without PMT (Experimental): Uterosacral Vaginal Vault Ligament Suspension (ULS) without Pelvic Muscle Training & Exercises (PMT)
  Interventions: Procedure: ULS

INTERVENTIONS:
Procedure: SSLF — sacrospinous ligament fixation (SSLF)
  Arms: SSLF and PMT; SSLF without PMT
Procedure: ULS — uterosacral vaginal vault ligament suspension (ULS)
  Arms: ULS and PMT; ULS without PMT
Behavioral: PMT — Pelvic muscle training and exercises (PMT)
  Arms: SSLF and PMT; ULS and PMT

SUMMARY:
Pelvic organ prolapse is common among women with a prevalence that has been estimated to be as high as 30%. Pelvic organ prolapse often involves a combination of support defects involving the anterior, posterior and/or apical vaginal segments. While the anterior vaginal wall is the segment most likely to demonstrate recurrent prolapse after reconstructive surgery, reoperations are highest among those who require apical suspension procedures with or without repair of other vaginal segments (12%-33%). Despite the substantial health impact, there is a paucity of high quality evidence to support different practices in the management of prolapse, particularly surgery. Thus, the objectives of the Operations and Pelvic Muscle Training in the Management of Apical Support Loss (OPTIMAL) Trial are:

1. to compare sacrospinous ligament fixation (SSLF) to uterosacral vaginal vault ligament suspension (ULS); and
2. to assess the role of perioperative behavioral therapy/pelvic muscle training (PMT) in women undergoing vaginal surgery for apical or uterine prolapse and stress urinary incontinence.

DETAILED DESCRIPTION:
Many women develop pelvic organ prolapse over the course of their lives. Pelvic organ prolapse is the downward descent of the pelvic organs (which include the uterus, bladder and bowel) into the vagina. Researchers estimate that between 7-10% of women will require surgery for prolapse sometime in their lifetime. Many will have more than one operation for the prolapse. Because this is such a common problem, the investigators in the Pelvic Floor Disorders Network strive to offer women the best treatment options. However, there were not enough carefully designed and conducted research studies to help guide them in this direction.

Women who are planning surgery for apical vaginal prolapse often experience bladder and bowel symptoms, as well as pressure and a bulge. These symptoms might include urinary leakage (urinary incontinence), urinary urgency (a sudden strong desire to urinate with fear that leakage may occur) or frequent urination, difficulty starting to urinate or perhaps a slow weak urinary stream, as well as accidental bowel leakage (fecal incontinence). After surgery, bladder and bowel symptoms may get better, get worse, or stay the same as before surgery. Sometimes new symptoms can start after surgery even if they weren't present before surgery.

The OPTIMAL study was designed to compare two commonly performed vaginal surgeries for pelvic organ prolapse. One is the sacrospinous ligament fixation, called SSLF for short. The other is the uterosacral ligament suspension, called ULS. Both surgeries involve attaching the top of the vagina, which has fallen down, to internal ligaments in the pelvis in order to resuspend the vagina and correct the prolapse.

The investigators were also interested in studying how the surgeries altered bladder and bowel symptoms. They had seen in other studies that behavioral and pelvic floor muscle therapy (PMT) is an effective therapy for stress and urge urinary incontinence, fecal incontinence, and other pelvic floor disorders. It is relatively easy to perform, and has rare side effects. They wondered if PMT around the time of surgery might further improve these symptoms.

The OPTIMAL study has two main purposes:

1. To find out which type of surgery, SSLF or ULS, has better results when used to repair prolapse of the top of the vagina,
2. To find out whether or not doing pelvic muscle exercises and behavioral changes around the time of surgery will affect both bladder and bowel symptoms after surgery, and the success of the prolapse repair.

Four Hundred women were enrolled into the OPTIMAL study, from January 2008 to May 2011. These women were randomly assigned to receive either the SSLF or the ULS surgery. They were randomly assigned to either receive the PMT training with a therapist before and after surgery or to not receive this therapy. So women fell into one of four groups:

1. SSLF plus PMT
2. ULS plus PMT
3. SSLF without PMT
4. ULS without PMT

Women in this study were followed closely at regular intervals for two years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Stage 2 to 4 prolapse
* Prolapse of the vaginal apex or cervix to at least half way into the vaginal canal (POPQ Point C > -TVL/2) [TVL stands for total vaginal length]
* Vaginal bulge symptoms as indicated by an affirmative response to either questions on the Pelvic Floor Distress Inventory (PFDI)
* Vaginal surgery for prolapse is planned, including a vaginal apical suspension procedure.
* Stress incontinence symptoms as indicated by an affirmative response to the PFDI Stress incontinence subscale
* Documentation of transurethral stress leakage on an office stress test or urodynamics with or without prolapse reduction within the previous 12 months
* A tension free vaginal tape (TVT) is planned to treat stress urinary incontinence.
* A pelvic muscle training (PMT) visit can be performed at least 2 weeks and not more than 4 weeks before surgery.
* Available for 24-months of follow-up.
* Able to complete study assessments, per clinician judgment
* Able and willing to provide written informed consent

Exclusion Criteria:

* Contraindication to sacrospinous ligament fixation (SSLF), uterosacral vaginal vault ligament suspension (ULS), or TVT in the opinion of the treating surgeon.
* History of previous surgery that included a SSLF or ULS. (Previous vaginal vault suspensions using other techniques or in which the previous technique is unknown are eligible.)
* Pelvic pain or dyspareunia due to levator ani spasm that would preclude a PMT program.
* History of previous synthetic sling procedure for stress incontinence.
* Previous adverse reaction to synthetic mesh.
* Urethral diverticulum, current or previous (i.e., repaired)
* History of femoral to femoral bypass.
* Current cytotoxic chemotherapy or current or history of pelvic radiation therapy.
* History of two inpatient hospitalizations for medical comorbidities in the previous 12 months.
* Subject wishes to retain her uterus. [Both ULS and SLS include removal of the uterus, if not previously removed]

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2008-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Barber, MD, Principal Investigator — The Cleveland Clinic
Locations (9):
- United States (9):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Kaiser Permanente Bellflower, Bellflower, California
  - University of California, San Diego Medical Center, La Jolla, California
  - Kaiser Permanente, San Diego, California
  - Loyola University Medical Center, Maywood, Illinois
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Texas Southwestern, Dallas, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barber MD, Brubaker L, Menefee S, Norton P, Borello-France D, Varner E, Schaffer J, Weidner A, Xu X, Spino C, Weber A; Pelvic Floor Disorders Network. Operations and pelvic muscle training in the management of apical support loss (OPTIMAL) trial: design and methods. Contemp Clin Trials. 2009 Mar;30(2):178-89. doi: 10.1016/j.cct.2008.12.001. Epub 2008 Dec 16. PMID 19130903
- [Derived] Borello-France D, Newman DK, Markland AD, Propst K, Jelovsek JE, Cichowski S, Gantz MG, Balgobin S, Jakus-Waldman S, Korbly N, Mazloomdoost D, Burgio KL; NICHD Pelvic Floor Disorders Network. Adherence to Perioperative Behavioral Therapy With Pelvic Floor Muscle Training in Women Receiving Vaginal Reconstructive Surgery for Pelvic Organ Prolapse. Phys Ther. 2023 Sep 1;103(9):pzad059. doi: 10.1093/ptj/pzad059. PMID 37318279
- [Derived] Jakus-Waldman S, Brubaker L, Jelovsek JE, Schaffer JI, Ellington DR, Mazloomdoost D, Whitworth R, Gantz MG; NICHD Pelvic Floor Disorders Network (PFDN). Risk Factors for Surgical Failure and Worsening Pelvic Floor Symptoms Within 5 Years After Vaginal Prolapse Repair. Obstet Gynecol. 2020 Nov;136(5):933-941. doi: 10.1097/AOG.0000000000004092. PMID 33030871
- [Derived] Lukacz ES, Sridhar A, Chermansky CJ, Rahn DD, Harvie HS, Gantz MG, Varner RE, Korbly NB, Mazloomdoost D; Eunice Kennedy Shriver National Institute of Child Health and Human Development Pelvic Floor Disorders Network (PFDN). Sexual Activity and Dyspareunia 1 Year After Surgical Repair of Pelvic Organ Prolapse. Obstet Gynecol. 2020 Sep;136(3):492-500. doi: 10.1097/AOG.0000000000003992. PMID 32769645
- [Derived] Sutkin G, Zyczynski HM, Sridhar A, Jelovsek JE, Rardin CR, Mazloomdoost D, Rahn DD, Nguyen JN, Andy UU, Meyer I, Gantz MG; NICHD Pelvic Floor Disorders Network. Association between adjuvant posterior repair and success of native tissue apical suspension. Am J Obstet Gynecol. 2020 Feb;222(2):161.e1-161.e8. doi: 10.1016/j.ajog.2019.08.024. Epub 2019 Aug 23. PMID 31449806
- [Derived] Lukacz ES, Warren LK, Richter HE, Brubaker L, Barber MD, Norton P, Weidner AC, Nguyen JN, Gantz MG. Quality of Life and Sexual Function 2 Years After Vaginal Surgery for Prolapse. Obstet Gynecol. 2016 Jun;127(6):1071-1079. doi: 10.1097/AOG.0000000000001442. PMID 27159758
- [Derived] Barber MD, Brubaker L, Burgio KL, Richter HE, Nygaard I, Weidner AC, Menefee SA, Lukacz ES, Norton P, Schaffer J, Nguyen JN, Borello-France D, Goode PS, Jakus-Waldman S, Spino C, Warren LK, Gantz MG, Meikle SF; Eunice Kennedy Shriver National Institute of Child Health and Human Development Pelvic Floor Disorders Network. Comparison of 2 transvaginal surgical approaches and perioperative behavioral therapy for apical vaginal prolapse: the OPTIMAL randomized trial. JAMA. 2014 Mar 12;311(10):1023-34. doi: 10.1001/jama.2014.1719. PMID 24618964
- [Derived] Barber MD, Kenton K, Janz NK, Hsu Y, Dyer KY, Greer WJ, White A, Meikle S, Ye W. Validation of the activities assessment scale in women undergoing pelvic reconstructive surgery. Female Pelvic Med Reconstr Surg. 2012 Jul-Aug;18(4):205-10. doi: 10.1097/SPV.0b013e31825e6422. PMID 22777368
- [Derived] Barber MD, Janz N, Kenton K, Hsu Y, Greer WJ, Dyer K, White A, Meikle S, Ye W. Validation of the surgical pain scales in women undergoing pelvic reconstructive surgery. Female Pelvic Med Reconstr Surg. 2012 Jul-Aug;18(4):198-204. doi: 10.1097/SPV.0b013e31825d65aa. PMID 22777367

RESULTS

PARTICIPANT FLOW:
Groups:
- SSLF+BPMT: Sacrospinous Ligament Fixation plus Perioperative Behavioral Therapy/Pelvic Muscle Training
- SSLF+USUAL: Sacrospinous Ligament Fixation plus No Perioperative Behavioral Therapy/Pelvic Muscle Training
- ULS+BPMT: Uterosacral Ligament Suspension plus Perioperative Behavioral Therapy/Pelvic Muscle Training
- ULS+USUAL: Uterosacral Ligament Suspension plus No Perioperative Behavioral Therapy/Pelvic Muscle Training
Period: Randomized to Surgical and BPMT Arms
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Started | 95 | 91 | 91 | 97
Completed | 95 | 91 | 91 | 97
Not Completed | 0 | 0 | 0 | 0
Period: Baseline to 6-Months
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Started | 95 | 91 | 91 | 97
Completed | 93 | 87 | 87 | 93
Not Completed | 2 | 4 | 4 | 4
Period: 6-Months to 24-Months
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Started | 93 | 87 | 87 | 93
Completed | 76 | 79 | 77 | 85
Not Completed | 17 | 8 | 10 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL | Total
Number analyzed (Participants) | 95 | 91 | 91 | 97 | 374
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (11.2) | 58.1 (10.7) | 58.7 (10.5) | 55.8 (11) | 57.2 (10.9)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 95 | 91 | 91 | 97 | 374
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 0 | 2
  Asian | 1 | 3 | 0 | 0 | 4
  Black or African American | 7 | 3 | 8 | 4 | 22
  Other | 6 | 7 | 9 | 9 | 31
  White | 80 | 77 | 74 | 84 | 315
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latina | 19 | 15 | 19 | 22 | 75
  Not Hispanic/Latina | 76 | 76 | 72 | 75 | 299
Insurance: Private/HMO [Count of Participants; unit: Participants]
  No | 33 | 30 | 28 | 32 | 123
  Yes | 62 | 61 | 63 | 65 | 251
Insurance: Medicare or Medicaid [Count of Participants; unit: Participants]
  No | 68 | 65 | 62 | 70 | 265
  Yes | 27 | 26 | 29 | 27 | 109
Insurance: Self-pay [Count of Participants; unit: Participants]
  No | 93 | 90 | 90 | 95 | 368
  Yes | 2 | 1 | 1 | 2 | 6
Insurance: Other [Count of Participants; unit: Participants]
  No | 77 | 74 | 76 | 75 | 302
  Yes | 18 | 17 | 15 | 22 | 72
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30 (6.2) | 28 (5.1) | 28.6 (4.9) | 28.8 (5.5) | 28.8 (5.5)
Current Smoker [Count of Participants; unit: Participants]
  No | 84 | 83 | 83 | 91 | 341
  Yes | 11 | 8 | 8 | 6 | 33
Diabetes [Count of Participants; unit: Participants]
  . | 5 | 2 | 0 | 1 | 8
  No | 78 | 81 | 76 | 87 | 322
  Yes | 12 | 8 | 15 | 9 | 44
Connective tissue disease [Count of Participants; unit: Participants]
  . | 1 | 1 | 0 | 3 | 5
  No | 93 | 90 | 90 | 91 | 364
  Yes | 1 | 0 | 1 | 3 | 5
Number of Vaginal Deliveries [Median (Full Range); unit: Number of deliveries] | 3 [0 to 8] | 2 [0 to 12] | 3 [0 to 15] | 3 [0 to 9] | 3 [0 to 15]
Number of Cesarean Deliveries [Median (Full Range); unit: Number of deliveries] | 0 [0 to 4] | 0 [0 to 2] | 0 [0 to 4] | 0 [0 to 2] | 0 [0 to 4]
Estrogen Use: Oral or patch [Count of Participants; unit: Participants]
  No | 84 | 76 | 80 | 88 | 328
  Yes | 11 | 15 | 11 | 9 | 46
Estrogen Use: Vaginal [Count of Participants; unit: Participants]
  No | 77 | 70 | 67 | 72 | 286
  Yes | 18 | 21 | 24 | 25 | 88
Menstrual Status [Count of Participants; unit: Participants]
  Not sure | 7 | 4 | 6 | 5 | 22
  Postmenopausal | 59 | 64 | 64 | 59 | 246
  Premenopausal | 29 | 23 | 21 | 33 | 106
Hysterectomy [Count of Participants; unit: Participants]
  No | 73 | 61 | 68 | 72 | 274
  Yes | 22 | 30 | 23 | 25 | 100
Prior Stress Urinary Incontinence Surgery [Count of Participants; unit: Participants]
  No | 93 | 87 | 87 | 94 | 361
  Yes | 2 | 4 | 4 | 3 | 13
Prior Pelvic Organ Prolapse Surgery [Count of Participants; unit: Participants]
  No | 89 | 80 | 88 | 91 | 348
  Yes | 6 | 11 | 3 | 6 | 26
Pelvic Organ Prolapse-Q stage [Count of Participants; unit: Participants] — The POP-Q assessment is a tool that measure the severity of prolapse. It measures nine points in the vagina with the hymen being the reference point. The distance to the reference point (in cm) is measured for the prolapsed and the severity stage is calculated. Higher stages indicate worse prolapse.
  Participants
    2 | 37 | 36 | 35 | 36 | 144
    3 | 54 | 48 | 51 | 59 | 212
    4 | 4 | 7 | 5 | 2 | 18

OUTCOME MEASURES:

1. Primary Outcome: Surgical Success
Description: The absence of the following: (1) descent of the vaginal apex more than one-third into the vaginal canal; (2) anterior or posterior vaginal wall descent beyond the hymen; (3) bothersome vaginal bulge symptoms as indicated by an affirmative response to either 'Do you usually have a sensation of bulging or protrusion from the vaginal area?' or 'Do you usually have a bulge or something falling out that you can see or feel in the vaginal area?' in the Pelvic Floor Distress Inventory and any response other than 'not at all' to the question 'How much does this bother you?'; or (4) re-treatment for prolapse by either surgery or pessary.
Time Frame: 24 months
Population: This outcome is analyzed in participants randomized to both surgical and behavioral interventions who had non-missing data for this 24-month outcome. There are minor differences between the Number of Participants Analyzed and the 24-month numbers in the Participant Flow module because of missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 72 | 77 | 73 | 82
Participants
  Failure | 25 | 30 | 28 | 27
  Success | 47 | 47 | 45 | 55

2. Primary Outcome: Anatomic Failure
Description: Anatomic failure is defined by one of the following: descent of the vaginal apex more than one-third into the vaginal canal, anterior or posterior vaginal wall descent beyond the hymen, or re-treatment for prolapse.
Time Frame: 24 months
Population: This outcome is analyzed in participants randomized to both surgical and behavioral interventions and who were in the study at 24 months.
Measure: Count of Participants; unit: Participants
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 76 | 79 | 77 | 85
Participants
  Failure | 18 | 23 | 19 | 19
  Non-failure | 58 | 56 | 58 | 66

3. Primary Outcome: Urinary Distress Inventory at 6 Months
Description: The Pelvic Floor Distress Inventory is a validated, self-reported instrument used to evaluate pelvic floor symptoms. It consists of 3 scales: 1. Pelvic Organ Prolapse Distress Inventory (POPDI, with 3 subscales), 2. Colorectal Anal Distress Inventory (CRADI, with 4 subscales), and 3. Urinary Distress Inventory (UDI, with 3 subscales). Scores are calculated by multiplying the mean value of all questions answered by 25 for the subscales and then adding the subscales. The range of responses for the UDI is: 0-300 with 0 (least distress) to 300 (most distress). Lower scores indicate better function / fewer symptoms.
Time Frame: 6 months
Population: This outcome is analyzed in participants randomized to both surgical and behavioral interventions who had non-missing data for this 6-month outcome. There are minor differences between the Number of Participants Analyzed and the 6-month numbers in the Participant Flow module because of missing data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 87 | 83 | 83 | 88
units on a scale | 30.6 [22.8 to 38.5] | 37.9 [27 to 48.8] | 27.4 [19.1 to 35.7] | 29.7 [21.3 to 38.1]

4. Secondary Outcome: Change From Baseline: Urinary Distress Inventory
Description: The Pelvic Floor Distress Inventory is a validated, self-reported instrument used to evaluate pelvic floor symptoms. It consists of 3 scales: 1. Pelvic Organ Prolapse Distress Inventory (POPDI, with 3 subscales), 2. Colorectal Anal Distress Inventory (CRADI, with 4 subscales), and 3. Urinary Distress Inventory (UDI, with 3 subscales). Scores are calculated by multiplying the mean value of all questions answered by 25 for the subscales and then adding the subscales. The range of responses for the UDI is: 0-300 with 0 (least distress) to 300 (most distress). Change = (24 Month Score - Baseline Score). Lower scores indicate better function / fewer symptoms.
Time Frame: Baseline and 24 months
Population: This outcome is analyzed in participants randomized to both surgical and behavioral interventions who had non-missing data for this 24-month outcome. There are differences between the Number of Participants Analyzed and the 24-month numbers in the Participant Flow module because of missing data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 76 | 72 | 70 | 74
units on a scale | -88.1 [-104.4 to -71.8] | -84.9 [-99.3 to -70.5] | -82.5 [-98.1 to -66.9] | -82.9 [-97 to -68.8]

5. Secondary Outcome: Change From Baseline: Pelvic Organ Prolapse Distress Inventory
Description: The Pelvic Floor Distress Inventory is a validated, self-reported instrument used to evaluate pelvic floor symptoms. It consists of 3 scales: 1. Pelvic Organ Prolapse Distress Inventory (POPDI, with 3 subscales), 2. Colorectal Anal Distress Inventory (CRADI, with 4 subscales), and 3. Urinary Distress Inventory (UDI, with 3 subscales). Scores are calculated by multiplying the mean value of all questions answered by 25 for the subscales and then adding the subscales. The range of responses for the POPDI is: 0-300 with 0 (least distress) to 300 (most distress). Change = (24 Month Score - Baseline Score). Lower scores indicate better function / fewer symptoms.
Time Frame: Baseline and 24 months
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 76 | 72 | 70 | 74
units on a scale | -77.4 [-93.7 to -61.1] | -70.6 [-87.9 to -53.4] | -79.3 [-96.6 to -62] | -66.4 [-80.8 to -52.1]

6. Secondary Outcome: Change From Baseline: Colorectal Anal Distress Inventory
Description: The Pelvic Floor Distress Inventory is a validated, self-reported instrument used to evaluate pelvic floor symptoms. It consists of 3 scales: 1. Pelvic Organ Prolapse Distress Inventory (POPDI, with 3 subscales), 2. Colorectal Anal Distress Inventory (CRADI, with 4 subscales), and 3. Urinary Distress Inventory (UDI, with 3 subscales). Scores are calculated by multiplying the mean value of all questions answered by 25 for the subscales and then adding the subscales. The range of responses for the CRADI is: 0-400 with 0 (least distress) to 400 (most distress). Change = (24 Month Score - Baseline Score). Lower scores indicate better function / fewer symptoms.
Time Frame: Baseline and 24 months
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 76 | 72 | 70 | 74
units on a scale | -48.6 [-68.9 to -28.2] | -46.5 [-66.1 to -26.8] | -61.4 [-78.6 to -44.2] | -52.4 [-70.2 to -34.7]

7. Secondary Outcome: Urinary Impact Questionnaire Change From Baseline to 24 Months
Description: The Pelvic Floor Impact Questionnaire measuring the impact of bladder, bowel, and vaginal symptoms on a woman's daily activities, relationships and emotions is composed of 3 scales: the Urinary Impact Questionnaire (UIQ; 4 subscales, range 0-400), the Pelvic Organ Prolapse Impact Questionnaire (POPIQ; 4 subscales, range 0-400), and the Colorectal-Anal Impact Questionnaire (CRAIQ; 4 subscales, range 0-400). Scores are calculated by multiplying the mean value of all answered questions for a subscale by 100 divided by 3. The subscales are then added together. The range of responses is: 0-400 with 0 (least negative impact) to 400 (most negative impact). Change = (24 Month Score - Baseline Score). Lower scores indicate better function / fewer symptoms.
Time Frame: Baseline and 24 months
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 76 | 72 | 70 | 74
units on a scale | -84 [-110.4 to -57.7] | -72.6 [-94.4 to -50.8] | -79 [-104.3 to -53.7] | -97.6 [-119.5 to -75.8]

8. Secondary Outcome: Pelvic Organ Prolapse Impact Questionnaire Change From Baseline to 24 Months
Description: The Pelvic Floor Impact Questionnaire measuring the impact of bladder, bowel, and vaginal symptoms on a woman's daily activities, relationships and emotions is composed of 3 scales: the Urinary Impact Questionnaire (UIQ; 4 subscales, range 0-400), the Pelvic Organ Prolapse Impact Questionnaire (POPIQ; 4 subscales, range 0-400), and the Colorectal-Anal Impact Questionnaire (CRAIQ; 4 subscales, range 0-400). Scores are calculated by multiplying the mean value of all answered questions for a subscale by 100 divided by 3. The subscales are then added together. The range of responses is: 0-400 with 0 (least negative impact) to 400 (most negative impact). Change = (Year 2 Score - Baseline Score). Lower scores indicate better function / fewer symptoms.
Time Frame: Baseline and 24 months
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 76 | 73 | 70 | 76
units on a scale | -67.5 [-94.6 to -40.4] | -49.1 [-70.9 to -27.3] | -59.4 [-86.1 to -32.6] | -82.2 [-103.7 to -60.7]

9. Secondary Outcome: Colorectal-Anal Impact Questionnaire Change From Baseline to 24 Months
Description: as for outcome 8
Time Frame: Baseline and 24 months
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 76 | 73 | 70 | 76
units on a scale | -40.9 [-67.8 to -14] | -21.6 [-41.8 to -1.4] | -29.2 [-54 to -4.3] | -42.5 [-60.7 to -24.2]

10. Secondary Outcome: Sexual Function 36 - Physical Health Component Score Change From Baseline to 24 Months
Description: Sexual Function 36 (SF36) - Physical Health Component Score is the physical health component of the Sexual Function 36 survey with scores ranging from 0 to 100 with higher scores meaning a better health state. Scales are scored according to the algorithm that describes the handling of the various types of questions included in the questionnaire. Several steps are involved in the scoring process: recoding items that require it; summing over items; and transforming raw scale scores to a 0 to 100 scale. This physical health component is a function of several constructs measured under the SF36: physical functioning, physical role, bodily pain, general health, and vitality.
Time Frame: Baseline and 24 months
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 75 | 71 | 71 | 75
units on a scale | 7.9 [5.3 to 10.4] | 4.8 [2.4 to 7.2] | 4.8 [2.6 to 6.9] | 6 [4 to 7.9]

11. Secondary Outcome: Sexual Function 36 - Mental Health Component Score Change From Baseline to 24 Months
Description: Sexual Function 36 (SF36) - Mental Health Component Score is the mental health component of the Sexual Function 36 survey with scores ranging from 0 to 100 with higher scores meaning a better health state. Scales are scored according to the algorithm that describes the handling of the various types of questions included in the questionnaire. Several steps are involved in the scoring process: recoding items that require it; summing over items; and transforming raw scale scores to a 0 to 100 scale.
Time Frame: Baseline and 24 months
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 75 | 71 | 71 | 75
units on a scale | 0.6 [-2.2 to 3.4] | 2 [-0.3 to 4.2] | 2.5 [0 to 5] | 1.1 [-1.7 to 4]

12. Secondary Outcome: Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire Change From Baseline to 24 Months
Description: Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ) is a survey of sexual functioning with scores ranging from 0 to 48 with higher scores meaning better sexual functioning. Patients were asked to answer 31 questions about their sexuality in the past 6 months.
Time Frame: Baseline and 24 months
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 35 | 25 | 27 | 37
units on a scale | 5.6 [3 to 8.2] | 4.6 [1.4 to 7.8] | 3.8 [0.9 to 6.6] | 6.6 [4.2 to 9.1]

ADVERSE EVENTS:
Time Frame: 24 Months
Arm/Group | ULS+BPMT | SSLF+BPMT | ULS+USUAL | SSLF+USUAL
Serious Adverse Events (participants affected / at risk) | 15/91 | 15/95 | 16/97 | 16/91
Other Adverse Events (participants affected / at risk) | 62/91 | 69/95 | 73/97 | 62/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ULS+BPMT (N=91) | SSLF+BPMT (N=95) | ULS+USUAL (N=97) | SSLF+USUAL (N=91)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hiatal Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal achalasia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suprapubic pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Unable to determine Preferred Term (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Biliary cholic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Allergic Reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Unable to determine Preferred Term (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PO2 decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Pain in Leg (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endometrial cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Transitonal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pudenal canal syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sciatic nerve neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression Suicidal (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast enlargement (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian vein thrombosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pelvic prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal Pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hiatus hernia (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Nephrectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prolapse repair (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ULS+BPMT (N=91) | SSLF+BPMT (N=95) | ULS+USUAL (N=97) | SSLF+USUAL (N=91)
OTHER ADVERSE EVENTS (General disorders) | 19 (19) | 21 (21) | 22 (22) | 25 (25)
MESH EROSION/EXPOSURE AT 4 WEEKS TO 24 MONTHS (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
SUTURE EXPOSURE AT 6 TO 24 MONTHS (General disorders) | 10 (10) | 18 (18) | 19 (19) | 14 (14)
BLADDER INJURY (Injury, poisoning and procedural complications) | 11 (11) | 10 (10) | 11 (11) | 8 (8)
BLOOD TRANSFUSION (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 5 (5) | 3 (3)
INTRAOPERTIVE URETERAL INJURY (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 4 (4) | 0 (0)
RECTAL INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TREATMENT - STENT PLACEMENT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TREATMENT - SUTURE REMOVED INTRAOPERATIVELY (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
URETERAL INJURY - DELAYED RECOGNITION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NEUROLOGIC PAIN REQUIRING TREATMENT (Nervous system disorders) | 8 (8) | 12 (12) | 5 (5) | 11 (11)
VAGINAL GRANULATION TISSUE AT 6 TO 24 MONTHS (Skin and subcutaneous tissue disorders) | 20 (20) | 17 (17) | 16 (16) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No